CLINICAL TRIAL: NCT06225102
Title: The Effect of Kegel Exercise on Menstruation Symptom, Severity of Dysmenorrheic Symptoms and Quality of Life in Nursing Students With Primary Dysmenorrhea: A Randomized Controlled Study
Brief Title: The Effect of Kegel Exercise in Nursing Students With Primary Dysmenorrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Özge PALANCI AY, RESEARCH ASSISTANT, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GU-SBF-OPA-01
Record Dates: First submitted 2024-01-13; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Primary Dysmenorrhea
Keywords: PRIMARY DYSMENORHEA; Kegel exercise; Nursing students; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The sample of the study consisted of 89 nursing students with primary dysmenorrhea (45 experimental group and 44 control group)
Who Masked: Participant
Masking Description: While it is known by the researchers that the students are in the experimental and control groups, it is not known by the students.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The intervention group was first given training on the definition of kegel exercises, diagnostic criteria, treatment, benefits and how to do kegel exercises on the Zoom platform.
  A second meeting was held for the participants of the initiative group who could not attend this training.
  At the same time, a message was sent to the WhatsApp application group where the intervention group was located three times a day by the researchers to remind them to do kegel exercises in the morning, noon and evening.
  Interventions: Behavioral: Kegel Exercise
- control group (No Intervention): No intervention was made in the control group

INTERVENTIONS:
Behavioral: Kegel Exercise — * Before teaching Kegel exercises, it was recommended that the person empty his bladder and wear comfortable clothing.
  * It was said that the person should extend his legs straight while exercising and not to contract his leg, hip and abdominal muscles and not to hold his breath while the pelvic floor muscles contract.
  * The relevant muscles were told to contract for 10 seconds and then relax for 10 seconds. The person was also asked to do the exercises during daily activities.
  * Exercise was implemented regularly 3 times a day (minimum 30-45 exercises) in the morning, noon and evening.
  Arms: experimental group

SUMMARY:
In this study, it was aimed to determine the effect of kegel exercise on menstruation symptoms, severity of dysmenorrheic symptoms and quality of life in nursing students with primary dysmenorrhea. The study was conducted as a single-blind randomized controlled trial.

DETAILED DESCRIPTION:
The study was conducted in a single-blind randomized controlled trial with 89 nursing students with primary dysmenorrhea. The experimental group was given kegel exercise training online, and after the training, a message was sent to remind them to do kegel exercises three times a day during the follow-up. No intervention was made in the control group.

Hypotheses of the Research

1. VAS total scores in interventions involving kegel exercise training and regular kegel exercise are lower than control interval rates (H1).
2. The total score of the Menstruation Symptom Scale within the participants who participated in kegel exercise training and regular kegel exercise was recorded, at lower rates than the distribution of control intervals (H1).
3. The Severity of Dysmenorrheic Symptoms in participants who participated in kegel exercise training and regular kegel exercise interventions were lower than the distribution of control intervals (H1).
4. The total scores of the Quality of Life Scale among those who participated in kegel exercise training and regular kegel exercises were higher than the proportions of the controlled rankings (H1).

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-25
* Giving 6 points or more to the least menstruation pain on the day that individuals experience the most severe dysmenorrhea symptoms (VAS) out of 10 points on the VAS Visual Pain Scale
* Being Nulliparous (never giving birth)
* Regular menstruation for the last six months
* Not having any gynecological diagnosis
* Not having had a gynecological operation
* Volunteering to participate in the study

Exclusion Criteria:

* Being a man
* Being married
* Being diagnosed with secondary dysmenorrhea
* Giving menstruation pain less than 6 points out of 10 on the VAS Visual Pain Scale.
* Taking painkillers 12 hours before the assessments.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | one week
  It was prepared in line with the literature. The form consists of a total of 25 questions, including information about socio-demographic information, pain during menstrual period, vaginal discharge characteristics, and practices regarding menstrual quantity.
Visual Analogue Scale | one week
  It was used to evaluate the pain intensity of individuals during their menstrual period.
  Individuals were asked to mark their pain level on a 10-centimeter (cm) horizontal line, meaning "0 (no pain)" and "10 (most severe pain)."
  Individuals responded by thinking about the pain they experienced during the first 3 days of their first, second, and third menstrual cycles.
The Menstrual Symptom Scale | Three months
  The scale consists of 22 items and is a five-point Likert type. Items 1-13 belong to "Negative effects/somatic complaints" sub-dimension, items 14-19 belong to "Menstrual pain symptoms" sub-dimension and items 20-22 belong to "Coping methods" sub-dimension. The Menstrual Symptom Scale score is calculated by averaging the total score of the items in the scale. Participants are asked to assign a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The scale has three sub-dimensions. The score obtained from the sub-dimensions is calculated by averaging the total score of the items in the sub-dimensions. An increase in the mean score for the sub-dimensions indicates an increase in the severity of menstrual symptoms related to that sub-dimension. Cronbach's Alpha value of the scale is 0.86
The Severity of Dysmenorrheic Symptoms | Three months
  The presence and magnitude of dysmenorrhoeic symptoms were assessed using this Likert-type scale (none = 0; mild = 1; moderate = 2; and severe = 3). The dimensions assessed by the scale are: Colicky pain in the lower abdomen, bloating, irritability, depression pain or tenderness in the breasts, back pain, gastrointestinal disorders headache, leg oedema
The Quality of Life Scale | Three months
  Item-total score correlations were calculated between 0.47-0.88. It is not possible to obtain a total score for the Short Form-36 quality of life scale. Instead, summary scores can be obtained for the physical and mental components of health in the Short Form-36 scale. Physical health components are physical function, physical role, pain and general health perception subscales, while mental health components are vitality, social function, emotional role and mental health subscales. In the summary scores, the lowest score is "0" and the highest score is "100" and a high score indicates good health status.

CONTACTS AND LOCATIONS:
Overall Officials: RUVEYDE AYDIN, Principal Investigator — Ondokuz Mayıs University; ÖZGE PALANCI AY, Principal Investigator — Gümüşhane Universıty; SONGÜL AKTAŞ, Principal Investigator — Karadeniz Technical University
Locations (1):
- Gümüşhane University, Faculty of Health Sciences, Department of Nursing, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No